CLINICAL TRIAL: NCT05180097
Title: A Randomized Phase II Study of Pembrolizumab and Brentuximab Vedotin Versus GDP, Followed by High Dose Chemotherapy and Autologous Stem Cell Transplantation for Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Pembrolizumab and Brentuximab Vedotin vs GDP and Stem Cell Transplant for Relapsed/Refractory Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD11
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Gemcitabine; Dexamethasone; Cisplatin; Brentuximab Vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDP (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin
- Brentuximab vedotin + Pembrolizumab (Active Comparator)
  Interventions: Drug: Brentuximab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 IV, 30 mins D1, D8
  Arms: GDP
Drug: Dexamethasone — 40mg daily PO, D1-D4
  Arms: GDP
Drug: Cisplatin — 75mg/m2 IV, 1 hour, D1
  Arms: GDP
Drug: Brentuximab vedotin — 1.8 mg/kg IV, 30 mins, Q21 days
  Arms: Brentuximab vedotin + Pembrolizumab
Drug: Pembrolizumab — 200mg IV, 30 mins, Q 21 days
  Arms: Brentuximab vedotin + Pembrolizumab

SUMMARY:
This study is being done to determine if two new drugs can shrink or eliminate classical Hodgkins lymphoma.

DETAILED DESCRIPTION:
Treatment given to participants whose disease has not responded to (refractory) or returned (relapsed) after previous treatment is known as salvage treatment.

The standard of care for participants who are not in a study is salvage treatment with gemcitabine, dexamethasone and cisplatin (GDP). This treatment can reduce symptoms and may stop the lymphoma from growing for a few months or longer. This standard treatment is approved by Health Canada

We are doing this study because we want to find out if treatment with Pembrolizumab and Brentuximab vedotin is better or worse than the standard of care for this type of cancer, classical Hodgkin lymphoma. The standard of care is defined as care most people get for your cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of classic Hodgkin lymphoma by histopathology and now have relapsed or refractory disease after anthracycline-containing chemotherapy and eligible for high dose chemotherapy and autologous stem cell transplant
* 18 years of age or greater
* ECOG performance status 0-1
* Clinically and/or radiologically measurable disease as per the Lugano 2014 classification
* Life expectancy > 90 days
* Absolute neutrophils ≥1.0 x 10^9/L; Platelets ≥75 x 10^9/L; Hemoglobin ≥80 g/L: Bilirubin ≤1.50 x UNL; AST and ALT ≤2.50 x UNL; Serum creatinine <1.55 x UNL or Creatinine clearance ≥30 mL/min
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires and/or health utility in either English or French
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Participants must be accessible for treatment and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of participant enrollment
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method during the study plus approximately 6 months after treatment completion
* All patients must have a tumour block from their primary diagnostic biopsy and relapse/refractory biopsy if available and the centre/pathologist must have agreed to release the block or recently cut slides for correlative analysis if the participant has consented. If the primary diagnostic biopsy is not accessible, the original pathology report should be submitted for review and a biopsy from the relapse/refractory disease must be submitted.

Exclusion Criteria:

* Participants who have received prior salvage systemic therapy for their relapsed or refractory disease.
* History of peripheral neuropathy or dyspnea ≥ grade 2
* Participants with a history of other malignancies except: adequately treated non-melanoma skin cancer and superficial bladder cancer, curatively treated in-situ cancer of the cervix or breast, or localized excised prostate cancer, other solid tumours curatively treated with no evidence of disease for > 3 years
* History of active CNS disease
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (at doses more than 10 mg prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first and any dose of trial treatment
* Has active autoimmune disease that has required systemic treatment in the past 3 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) or history of allogeneic transplantation. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of human immunodeficiency virus (HIV), active Hepatitis C Virus infection, active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Participants that are Hepatitis B core antibody positive are eligible if they are HBV DNA negative and are concurrently treated with anti-viral therapy. Participants with a past history of hepatitis C who have eradicated the virus are eligible
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, angina, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Documented history of cerebral vascular event (stroke or transient ischemic attack)
* History of progressive multifocal leukoencephalopathy (PML).
* Any serious active disease or co-morbid medical condition, including psychiatric illness, judged by the local investigator to preclude safe administration of the planned protocol treatment or required follow-up
* Any other serious intercurrent illness, life-threatening condition, organ system dysfunction, or medical condition judged by the local investigator to compromise the subject's safety (for example): active, uncontrolled bacterial, fungal or viral infection; clinically significant cardiac dysfunction or cardiovascular disease
* Participants who have been vaccinated with live, attenuated vaccines within 4 weeks of enrollment
* Pregnant or lactating females, or women/men of childbearing potential not willing to use an adequate method of birth control for the duration of the study through 6 months after the last dose of trial treatment
* Participants are not eligible if they have had a prior infusion reaction to the study drugs or their components > grade 2
* Participant has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Participant has had an allogenic tissue/solid organ transplant
* Concurrent or within the previous 4 weeks of randomization, treatment with other investigational drugs or anti-cancer therapy
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A one-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate by PET Deauville criteria (score 1-3) of pembrolizumab and brentuximab vedotin compared to standard GDP (gemcitabine, dexamethasone, cisplatin) given as salvage therapy | 52 months

SECONDARY OUTCOMES:
Progression-free survival | 52 months
Event-free survival | 52 months
Overall survival | 52 months
Successful stem cell collection rate | 52 months
Transplantation rate | 52 months
Number and severity of adverse events | 52 months
Participant-reported Quality of Life utilizing EORTC QLQ-C30 | 52 months
Participant-reported toxicity utilizing PRO-CTCAE | 52 months
Participant-reported Quality of Life utilizing FACT-LYM evaluating symptoms and concerns associated specifically with the lymphoma disease and/or disease treatment. | 52 months
Participant-reported Quality of Life utilizing FACT/GOG-Ntx-Subscale specifically with chemotherapy-induced neuropathy | 52 months
Health Economics utilizing EQ-5D-5L | 52 months
Health Economics financial toxicity utilizing FACIT-COST | 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Savage, Study Chair — BCCA-Vancouver Cancer Centre; John Kuruvilla, Study Chair — University Health Network, Princess Margaret Hospital
Locations (18):
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Shoalhaven Cancer Care Centre, Nowra, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Canada (12):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA - Vancouver, Vancouver, British Columbia
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No